CLINICAL TRIAL: NCT06166459
Title: Drug-coated Balloon Combined With Provisional Drug-eluting Stent Implantation (Yao Strategy) for the Treatment of de Novo Medina 0,1,0 or 0,0,1 Bifurcation Lesion
Brief Title: Yao Strategy for the Treatment of de Novo Medina 0,1,0 or 0,0,1 Bifurcation Lesion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Third People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-02-022-K01
Record Dates: First submitted 2023-12-03; First posted 2023-12-12 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease; Bifurcation Lesion
Keywords: drug-coated balloon; percutaneous coronary intervention; drug-eluting stent; Yao strategy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yao technique (Experimental): The following 2 treatment strategies are available. (1) DCB combined with provisional DES implantation 1-2 mm distally to the lesion ostium whenever this was required (DCB+pDES strategy). (2) DES implantation 1-2 mm distally to the lesion ostium followed by DCB (DES+DCB strategy).
  Interventions: Procedure: Drug-coated balloon combined with provisional drug-eluting stent implantation

INTERVENTIONS:
Procedure: Drug-coated balloon combined with provisional drug-eluting stent implantation — (1) DCB combined with provisional DES implantation 1-2 mm distally to the ostium lesion whenever this was required (DCB+pDES strategy). (2) DES implantation 1-2 mm distally to the ostium lesions followed by DCB treatment (DES+DCB strategy).

SUMMARY:
Percutaneous coronary intervention for coronary bifurcation lesions represents one of the most challenging procedures in interventional cardiology because of lower angiographic success rate and increased risk of procedural complications. The study is designed to enroll 200 patients with acute or chronic coronary syndromes that meet the indications for intervention and with angiographic confirmed de novo Medina type 0,1,0 or 0,0,1 bifurcation lesion. In view of the potential risks of using DCB alone in the treatment of de novo bifurcation lesions, the following 2 treatment strategies are available. (1) DCB combined with provisional DES implantation 1-2 mm distally to the lesion ostium whenever this was required (DCB+pDES strategy). (2) DES implantation 1-2 mm distally to the lesion ostium followed by DCB (DES+DCB strategy). The primary endpoint was late lumen loss and major adverse cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects at the age between ≥18 and ≤80 years old;
2. De novo native lesion, Median type 010/001 bifurcation lesion;
3. The reference diameter of the target vessel was 2.75-4.0mm and the length was less than 40mm;
4. Subjects are willing to participate in the study, sign informed consent form, and accept clinical follow-up.

Exclusion Criteria:

1. The diameter stenosis of adjacent branch vessel ostium ≥50%;
2. Acute ST-segment elevation myocardial infarction;
3. Stents implanted within 10 mm proximal or distal to the target lesion;
4. Aneurysm within 10 mm proximal or distal to the target lesion;
5. There is target vessel distortion or severe calcification lesion, so balloon catheter fails to pass;
6. Previous coronary artery bypass grafting;
7. Evidence for extensive thrombus within target vessel;
8. Evidence of heart failure by at least one of the following: a. Most recent LVEF ≤35%, or b. Current heart failure defined as dyspnea at rest (NYHA class IV assessed day of procedure), or c. Killip class ≥2 (post STEMI patients);
9. Subjects with a life expectancy of ≤1 year;
10. Subjects with stroke, peptic ulcer, or gastrointestinal bleeding within the past 6 months;
11. Subjects with severe renal failure (eGFR<30ml/minute), failure to comply with angiography conditions;
12. Subjects who are intolerance to aspirin and/or clopidogrel or ticagrelor or have contraindications;
13. Subjects who are intolerance or allergic to heparin, contrast agent;
14. Patients who are participating in the clinical trial of other drug or device without reaching the time limit of primary endpoint;
15. Subjects who are not applicable to be enrolled by investigators due to other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-22 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
late lumen loss | 9 months follow-up
  post-procedural minimum lumen diameter minus follow-up minimum lumen diameter.
major adverse cardiovascular events | 1 year
  include cardiac death, non-fatal myocardial infarction, and target lesion revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Yaojun Zhang, Dr, Study Chair — Xuzhou Third People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Escarcega RO. What is the Optimal Technique for Ostial Left Anterior Descending Artery Lesions? Cardiovasc Revasc Med. 2019 Dec;20(12):1063-1064. doi: 10.1016/j.carrev.2019.10.003. Epub 2019 Oct 22. No abstract available. PMID 31669112
- [Background] Dishmon DA, Elhaddi A, Packard K, Gupta V, Fischell TA. High incidence of inaccurate stent placement in the treatment of coronary aorto-ostial disease. J Invasive Cardiol. 2011 Aug;23(8):322-6. PMID 21828393
- [Background] Hildick-Smith DJ, Shapiro LM. Ostial left anterior descending coronary artery stent positioning: partial preinflation prevents stent oscillation and facilitates accurate deployment. J Interv Cardiol. 2001 Aug;14(4):439-42. doi: 10.1111/j.1540-8183.2001.tb00355.x. PMID 12053499
- [Background] Cayli M, Elbasan Z, Gur M, Seker T, Ucar H, Kuloglu O, Sen O, Sahin DY, Kalkan GY. Modified flower petal technique in the treatment of Medina type 0,0,1 or 0,1,0 lesions. EuroIntervention. 2015 Nov;11(7):772-9. doi: 10.4244/EIJV11I7A154. PMID 26603986
- [Background] Gutierrez-Chico JL, Villanueva-Benito I, Villanueva-Montoto L, Vazquez-Fernandez S, Kleinecke C, Gielen S, Iniguez-Romo A. Szabo technique versus conventional angiographic placement in bifurcations 010-001 of Medina and in aorto-ostial stenting: angiographic and procedural results. EuroIntervention. 2010 Feb;5(7):801-8. doi: 10.4244/eijv5i7a134. PMID 20142194
- [Background] Chen GC, Lu XM, Song YM, Gyawail L, Geng ZH, Song MB, Qian DH, Zhang YP, Ni DC, He Y. A 3-year experience of a simple, novel technique for accurate ostial/non-ostial coronary stenting: The buddy balloon anchor stent technique. Catheter Cardiovasc Interv. 2018 Nov 15;92(6):1147-1152. doi: 10.1002/ccd.27667. Epub 2018 Jul 18. PMID 30019847
- [Background] Yang ZK, Hu J, Ding FH, Ni JW, Zhang RY, Shen WF. One-year outcome of single-stent crossover versus accurate ostial stenting for isolated left anterior descending ostial stenosis. Coron Artery Dis. 2022 Jan 1;31(1):e67-e72. doi: 10.1097/MCA.0000000000001071. PMID 34010192
- [Background] Elkhateeb O, Thambi S, Beydoun H, Bishop H, Quraishi A, Kidwai B, Title L. Long-term outcomes following ostial left anterior descending artery intervention with or without crossover to left-main. Am J Cardiovasc Dis. 2022 Apr 15;12(2):73-80. eCollection 2022. PMID 35600287
- [Background] Vaquerizo B, Fernandez-Nofreiras E, Oategui I, Suarez de Lezo J, Rumoroso JR, Martin P, Routledge H, Tizon-Marcos H. Second-Generation Drug-Eluting Balloon for Ostial Side Branch Lesions (001-Bifurcations): Mid-Term Clinical and Angiographic Results. J Interv Cardiol. 2016 Jun;29(3):285-92. doi: 10.1111/joic.12292. PMID 27245124
- [Background] Erdogan E, Li Z, Zhu YX, Tufaro V, Feng SL, Li Q, Liang L, Chang S, Bu LT, Liu B, Zhou QH, Yap NAL, Bourantas CV, Zhang YJ. DCB combined with provisional DES implantation in the treatment of De Novo Medina 0,1,0 or 0,0,1 left main coronary bifurcation lesions: A proof-of-concept study. Anatol J Cardiol. 2022 Mar;26(3):218-225. doi: 10.5152/AnatolJCardiol.2021.1157. PMID 35346908